CLINICAL TRIAL: NCT06535763
Title: Impact and Influence of the Use of Hypnosis Adapted to People With Severe Stage Neurocognitive Disorder (HAPNeSS) on the Professional Practices of EHPAD (Establishment for Dependent Elderly People) Caregivers With Elderly Residents
Acronym: HAPNeSS-E
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/87
Record Dates: First submitted 2024-07-23; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease; Behavior Disorders
Keywords: self-hypnosis; formation; seniors
MeSH Terms: conditions — Alzheimer Disease; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- professional caregiver: nurse, care assistant, gerontological care assistant, psychologist, coordinating doctor, psychomotrician, occupational therapist in one of the 3 EHPADs in the study
  Interventions: Other: professional caregiver

INTERVENTIONS:
Other: professional caregiver — Care professionals will be questioned using a self-administered Quality of Life at Work scale, as well as a second scale (before and after training, with one test per day for 3 consecutive working days) asking about the number of work situations involving behavioral disorders in the residents under their care, and how they use the HAPNeSS method to deal with these situations.
  The effects of the HAPNeSS method on caregivers' professional practices (actions taken, performance of tasks, relations with residents, etc.) and their feelings on the subject, will be collected in two semi-structured interviews (with half the participants selected at random) conducted before and after the training course by the research team's occupational psychologist.

SUMMARY:
The aim of this study is to propose a non-anxiety-inducing method of managing behavioral disorders for patients and healthcare professionals. The main objective of this study is to evaluate the implementation, use and effects of HAPNeSS (Hypnosis Adapted to People with Severe Neurocognitive Disorders) training on the management of residents aged over 75 with moderately severe to severe Alzheimer's disease or a related disorder, who may present behavioral disorders, with caregivers working in EHPAD.

DETAILED DESCRIPTION:
The HAPNeSS method would offer caregivers the opportunity to find solutions to difficulties encountered (behavioral disorders, difficult care, etc.), to move away from pure technicality to reinvest in the relationship with the patient, and to find soothing, respectful and benevolent channels of communication. The aim of this study is to evaluate the effects of HAPNeSS (Hypnosis Adapted to People with Severe Neurocognitive Disorders) training on the care of residents over 75 with moderately severe to severe Alzheimer's disease or related disorders, who may present behavioral problems.

But also to measure, within each establishment, the effects of the HAPNeSS method, on the professional practices of caregivers (actions implemented, execution of missions, relationship with residents...) and to gather their feelings. These objectives therefore aim to collect and evaluate the effects of this method on the relationship between patients and caregivers, as well as on the latter's QWL. To achieve this, the research team organized 4 visits to the EHPADs participating in the study, spread over 6 months. Training takes place over 3 and then 2 days. Before and after the training, a visit at the beginning and end of the study will enable the scales to be administered and the interviews to be conducted. The data collected will be the subject of a mixed statistical analysis. Throughout the study, the research team will monitor the learning and development of each care professional.

ELIGIBILITY:
Inclusion Criteria:

EHPAD staff meeting the following criteria will be included in the study:

* Nurses, care assistants, gerontological care assistants, psychologists, coordinating physicians, psychomotor therapists, occupational therapists;
* More than one year's experience in the structure.

The study will examine the individual perceptions of EHPAD professionals of patients meeting the following criteria:

* Be a resident of an EHPAD ;
* suffering from a moderately severe or severe major neurocognitive disorder;
* over 75 years of age.

Exclusion Criteria:

EHPAD professionals will not be included:

* Not fluent in French,
* Not wishing to be trained in hypnosis.

The individual perception of EHPAD professionals of patients meeting these criteria will not be questioned in the study:

* Minor neurocognitive impairment, major neurocognitive impairment at a mild or moderate stage, or no cognitive impairment;
* under 75 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: EHPAD staff meeting :
  * Nurses, care assistants, gerontological care assistants, psychologists, coordinating physicians, psychomotor therapists, occupational therapists; with more than one year's experience in the structure.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Impact of HAPNeSS on the management of work situations involving behavioral disorders. | Month 2 and month 6
  Number of work situations which the carer feels he/she has had difficulty managing, involving a resident with a neurocognitive disorder and behavioural problems.

SECONDARY OUTCOMES:
Effects of HAPNeSS method to professional practices | Month 2 and month 6
  Scale QENA, minimum value 69 and maximum value 276. Analysis of feelings and impressions of professionals will be obtained from the analysis of the semi-directed interviews (qualitative analysis).

CONTACTS AND LOCATIONS:
Overall Officials: Marie FLOCCIA, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Chu de Bordeaux, Pessac, France

IPD SHARING:
Plan to Share IPD: No